CLINICAL TRIAL: NCT01396213
Title: A Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Different Doses of Larazotide Acetate for the Treatment of Celiac Disease
Brief Title: A Double-blind Placebo-controlled Study to Evaluate Larazotide Acetate for the Treatment of Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clin1001-012
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
Keywords: larazotide acetate
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Larazotide Acetate 0.5 mg (Experimental): larazotide acetate 0.5 mg capsules TID
  Interventions: Drug: Larazotide Acetate
- Larazotide Acetate 1 mg (Experimental): larazotide acetate 1 mg capsules TID
  Interventions: Drug: Larazotide Acetate
- Larazotide Acetate 2 mg (Experimental): larazotide acetate 2 mg capsules TID
  Interventions: Drug: Larazotide Acetate
- Placebo (Placebo Comparator): placebo capsules TID
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Larazotide Acetate — gelatin capsule
  Other Names: AT-1001; INN-202
  Arms: Larazotide Acetate 0.5 mg; Larazotide Acetate 1 mg; Larazotide Acetate 2 mg
Drug: placebo — gelatin capsule
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled Phase 2B study to evaluate the efficacy and safety of Larazotide Acetate in the treatment of patients with celiac disease who have persistent symptoms despite being on a gluten-free diet.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled Phase 2B study to evaluate the efficacy and safety of three different doses (0.5, 1 and 2 mg TID) of Larazotide Acetate as an adjunct to gluten-free diet in the treatment of patients with celiac disease (CD). The diagnosis of CD must have been established by jejunal biopsy as well as serology at some point in time prior to entry into the study. Patients must have symptoms despite being on a gluten-free diet as defined by a celiac disease domain of the gastrointestinal symptoms rating scale equal to or more than 2.0.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with biopsy proven and serology-confirmed celiac disease on a gluten-free diet for at least 12 months
* measurable serology at screening
* CeD GSRS score of ≥ 2.0 prior to randomization
* experiencing symptoms (ie, diarrhea, abdominal pain, bloating, nausea, or stomachache)
* willing to maintain current diet gluten-free diet throughout the duration of the study.

Exclusion Criteria:

* refractory celiac disease or severe complications of celiac disease (eg, EATL, ulcerative jejunitis, perforation, etc.)
* chronic active GI disease other than celiac disease
* diabetes (Type 1 or 2) or other autoimmune disease that might interfere with the conduct of the study
* hemoglobin value < 8.5 g/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2013-08-20 (Actual); Study Completion 2013-08-20 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of larazotide acetate versus placebo for the treatment of celiac disease in adults as an adjunct to a gluten-free diet | CeD GSRS was completed weekly Baseline through the end of 12-week double-blind treatment period.
  The primary efficacy endpoint was average on-treatment (Baseline to Week 12) score of theCeliac Disease Gastrointestinal Symptom Rating Scale (CeD GSRS).

SECONDARY OUTCOMES:
Assess the safety and tolerability of larazotide acetate in subjects with active celiac disease | Up to 12 weeks
  Safety endpoints assessed in this study were adverse events, vital signs, physical examination results, clinical laboratory test results, concomitant medication usage and ECG results
Validate a CeD PRO diary instrument in subjects with celiac disease | The CeD PRO was administered daily throughout the study.
  The CeD PRO is a 12-item questionnaire that was developed to assess symptom severity in clinical trials in subjects with celiac disease. Items in the questionnaire were formulated based on one-on-one interviews with subjects with celiac disease and thus reflect the symptoms that subjects consider part of their celiac disease experience. Subjects rated their symptom severity on an 11-point (0-10) scale. Symptoms included abdominal cramping, abdominal pain, bloating, constipation, diarrhea, gas, loose stools, nausea, vomiting, headache, and tiredness. The questionnaire was designed as a self-administered daily diary, to be completed at the same time each day, and required < 10 minutes to complete.
Compare various efficacy endpoints during 12 weeks of double-blind treatment | GSRS - weekly; BSFS - daily; CGA - screening, baseline, Week 12 and follow-up visits; CeD-QoL and SF12v2 - start of placebo run-in, Week 12 and follow-up visits; CD and CFDCQ - follow-up visit.
  Additional efficacy assessments comprised a variety of known scales used for evaluating subjects with celiac disease, including the Gastrointestinal Symptoms Rating Scale (GSRS), Bristol Stool Form Scale (BSFS), Short Form 12 health survey Version 2 (SF12v2), Celiac Disease Quality of Life (CeD-QoL) scale, and the Clinical Global Assessment (CGA). A Gluten-Free Diet Compliance Questionnaire (GFDCQ) and Celiac Dietary Adherence Test (CDAT) were also included to assess compliance with the gluten-free diet.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Director — Sponsor GmbH
Locations (61):
- United States (55):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Tucson, Arizona
  - Oceanside, California
  - Orange, California
  - San Francisco, California
  - Santa Monica, California
  - Walnut Creek, California
  - Denver, Colorado
  - Boynton Beach, Florida
  - Edgewater, Florida
  - Orlando, Florida
  - Summerfield, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Rockford, Illinois
  - West Des Moines, Iowa
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Chesterfield, Michigan
  - Wyoming, Michigan
  - Duluth, Minnesota
  - Rochester, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Missoula, Montana
  - Las Vegas, Nevada
  - Marlton, New Jersey
  - Lake Success, New York
  - New York, New York
  - Rochester, New York
  - Cary, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Mentor, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Perkasie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Chattanooga, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - St. George, Utah
  - Alexandria, Virginia
  - Charlottesville, Virginia
  - Seattle, Washington
- Canada (6):
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leffler DA, Kelly CP, Green PH, Fedorak RN, DiMarino A, Perrow W, Rasmussen H, Wang C, Bercik P, Bachir NM, Murray JA. Larazotide acetate for persistent symptoms of celiac disease despite a gluten-free diet: a randomized controlled trial. Gastroenterology. 2015 Jun;148(7):1311-9.e6. doi: 10.1053/j.gastro.2015.02.008. Epub 2015 Feb 13. PMID 25683116